CLINICAL TRIAL: NCT00375934
Title: Multicenter Study to Evaluate the Analgesic Efficacy of XP21L in Subjects With Pain Following Bunionectomy Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xanodyne Pharmaceuticals (Industry)
Responsible Party: Gary Shangold, M.D. / Chief Medical Officer, Xanodyne Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XP21L-302
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-05

CONDITIONS: Pain, Postoperative
Keywords: Bunionectomy; Bunion surgery; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Diclofenac

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: diclofenac potassium (XP21L)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: diclofenac potassium (XP21L) — 25 mg capsule, every 6 hours
  Other Names: Zipsor Liquid Filled Capsule; XP21L
  Arms: 1
Drug: Placebo — Oral placebo capsule, every 6 hours
  Arms: 2

SUMMARY:
A multicenter study to evaluate the analgesic efficacy of XP21L in subjects with pain following bunionectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Have undergone bunionectomy surgery
* Have achieved adequate post-surgical pain

Exclusion Criteria:

* Confounding medical conditions which preclude study participation
* Participated in a study of another investigational drug or device within 30 days prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-09; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Investigative Site, Austin, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, San Marcos, Texas
  - Investigative Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Daniels SE, Riff D, Diamond E, Clark F, Boesing SE. An assessment of the efficacy and safety of diclofenac potassium liquid-filled capsules in patients with various levels of baseline pain intensity. Curr Med Res Opin. 2012 Jun;28(6):953-61. doi: 10.1185/03007995.2012.694363. Epub 2012 Jun 11. PMID 22587481
- [Derived] Daniels SE, Baum DR, Clark F, Golf MH, McDonnell ME, Boesing SE. Diclofenac potassium liquid-filled soft gelatin capsules for the treatment of postbunionectomy pain. Curr Med Res Opin. 2010 Oct;26(10):2375-84. doi: 10.1185/03007995.2010.515478. PMID 20804444
- See also: Related Info — http://www.zipsor.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Zipsor (Diclofenac Potassium) Liquid Filled Capsule: 25 mg capsule, every 6 hours
Period: Overall Study
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Started | 99 | 101
Completed | 96 | 95
Not Completed | 3 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo | Total
Number analyzed (Participants) | 99 | 101 | 200
Age Continuous [Mean (Standard Deviation); unit: years] | 41 (13) | 40 (12) | 40 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 172
  Male | 13 | 15 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 66 | 57 | 123
  Black | 8 | 15 | 23
  Asian | 2 | 2 | 4
  Hispanic | 21 | 26 | 47
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 99 | 101 | 200
Baseline Pain Score [Mean (Standard Deviation); unit: units on a scale] — Pain intensity scores were measured using an 11-point numerical pain rating scale (NPRS) with 0=no pain to 10=worst possible pain
  units on a scale | 7.5 (1.6) | 7.4 (1.4) | 7.5 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Average Numeric Pain Rating Score (NPRS) Over 48 Hours After Bunionectomy
Description: Pain intensity scores were measured using an 11-point numerical pain rating scale (NPRS) with 0=no pain to 10=worst possible pain
Time Frame: Over 48 hours after bunionectomy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 99 | 101
units on a scale | 3.3 (2.2) | 5.7 (2.1)

2. Secondary Outcome: Number of Patients With Perceptible Pain Relief on Day 1
Description: Times to onset of Perceptible and Meaningful Relief were determined using the double-stopwatch method.
Time Frame: 8 hours post single dose
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 99 | 101
participants | 72 | 63

3. Secondary Outcome: Median Time to Onset of Pain Relief in Patients With Perceptible Pain Relief on Day 1
Time Frame: 8 hours post single dose
Population: Number of participants analyzed includes only the number of participants with perceptible pain relief on Day 1 (see previous outcome measure #2).
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 72 | 63
minutes | 42.9 [33.6 to 53.3] | 36.0 [29.8 to 60.4]

4. Secondary Outcome: Number of Patients With Meaningful Pain Relief on Day 1
Description: Times to onset of Perceptible and Meaningful Relief were determined using the double-stopwatch method.
Time Frame: 8 hours post single dose
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 99 | 101
participants | 50 | 30

5. Secondary Outcome: Median Time to Onset of Pain Relief in Patients With Meaningful Pain Relief on Day 1
Time Frame: 8 hours post single dose
Population: Number of participants analyzed includes only the number of participants with meaningful pain relief on Day 1 (see previous outcome measure #4).
  Number of patients in the placebo group is intentionally blank as the data (eg., median and upper CI) were not calculable (see post-hoc outcome measure #12 for available placebo results).
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 50 | 0
minutes | 90.6 [85.0 to 119.7] |

6. Secondary Outcome: Total Pain Relief (TOTPAR) Scores 8 Hours Post Initial Dose of Study Drug
Description: Pain relief was rated using a 5-point categorial scale (0=none, 1=a little, 2=some, 3=a lot, and 4=complete) at time of dose (time=0) and over 15 time points afterwards (10, 15, 20, 30, 45, and 60 minutes and at 1.5, 2, 2.5, 3, 4, 5, 6, 7, and 8 hours after the initial dose on Day 1 or until time of re-medication). A score of 0 across all time points would be the lowest (worst) and a score of 60 (4 X 15 time points) would be the highest (best) possible score.
Time Frame: 8 hourse post single dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 99 | 101
units on a scale | 5.9 (7.4) | 1.9 (3.6)

7. Secondary Outcome: Number of Patients With at Least 30% Reduction in Pain Intensity After First Dose of Study Drug
Time Frame: 8 hours post single dose
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 99 | 101
participants | 51 | 31

8. Secondary Outcome: Time to Onset of at Least 30% Reduction in Pain Intensity After First Dose of Study Drug
Time Frame: 8 hours post single dose
Population: Number of participants analyzed includes only the number of participants with at least 30% reduction in pain intensity after first dose of study drug (see previous outcome measure #7).
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 51 | 31
minutes | 110 [90 to 147] | 300 [120 to 300]

9. Secondary Outcome: Number of Patients Who Required Rescue Medication on Day 1
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 99 | 101
participants | 53 | 93

10. Secondary Outcome: Number of Patients Who Required Rescue Medication on Day 2
Time Frame: Day 2
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 99 | 101
participants | 30 | 68

11. Secondary Outcome: Number of Patients Who Required Rescue Medication on Day 3
Description: Day 3 data reflect the use of rescue medication only up to the time of discharge.
Time Frame: Day 3
Measure: Number; unit: participants
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Number analyzed (Participants) | 99 | 101
participants | 4 | 19

ADVERSE EVENTS:
Arm/Group | Zipsor (Diclofenac Potassium) Liquid Filled Capsule | Placebo
Serious Adverse Events (participants affected / at risk) | 0/99 | 1/101
Other Adverse Events (participants affected / at risk) | 46/99 | 63/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zipsor (Diclofenac Potassium) Liquid Filled Capsule (N=99) | Placebo (N=101)
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zipsor (Diclofenac Potassium) Liquid Filled Capsule (N=99) | Placebo (N=101)
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 4 | 5
Diarrhea (Gastrointestinal disorders) | 0 | 3
Dry Mouth (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 18 | 27
Vomiting (Gastrointestinal disorders) | 8 | 8
Feeling Hot (General disorders) | 0 | 3
Injection site pain (General disorders) | 0 | 3
Alanine aminotransferase increased (Investigations) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 6 | 8
Headache (Nervous system disorders) | 7 | 7
Somnolence (Nervous system disorders) | 6 | 5
Nightmare (Psychiatric disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other